CLINICAL TRIAL: NCT05637593
Title: Effects of Training Involving Rhythmic Auditory Stimulation on Upper-limb Movements in Patients With Parkinson's Disease
Brief Title: Rhythmic Auditory Stimulation on Upper-limb Movements in PD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, FAN Wei, PhD Student, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HongKongPU21037721r_20221117
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Acoustic Stimulation; Parkinson Disease; Movement, Abnormal; Bradykinesia; Arm
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Hypokinesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the RAS group (Experimental): The RAS group will receive upper-limb movement training with the aid of RAS;
  Interventions: Behavioral: Upper-limb movement training with the aid of RAS
- the no-RAS group (Active Comparator): The no-RAS group will receive upper-limb movement training without the aid of RAS.
  Interventions: Behavioral: Upper-limb movement training without the aid of RAS

INTERVENTIONS:
Behavioral: Upper-limb movement training with the aid of RAS — Three target bowls, labeled as the left, middle, and right target bowl, will be placed on the table at an equal distance from the main bowl. The distance between a target bowl and the main bowl is set at 30 cm. Wooden beads with a diameter of 2 cm will be put in target bowls. The main bowl will be placed in front of the patient.
  Patients will be asked to listen to the RAS sound, use the right hand to take one bead at a time from the left target bowl to the main bowl, repeat this movement for the middle and right target bowls, and keep repeating this order. They should keep their movements consistent with the sound of the RAS, with one RAS sound corresponding to one pick-up movement.
  Each daily training will consist of three rounds separated by two 5-minute breaks. Each round will consist of four consecutive sessions (for each session: 2-minute training followed by a 30-second break). The training will last for a total of 21 days.
  Arms: the RAS group
Behavioral: Upper-limb movement training without the aid of RAS — Three target bowls, labeled as the left, middle, and right target bowl, will be placed on the table at an equal distance from the main bowl. The distance between a target bowl and the main bowl is set at 30 cm. Wooden beads with a diameter of 2 cm will be put in target bowls. The main bowl will be placed in front of the patient.
  Patients will be asked to use the right hand to take one bead at a time from the left target bowl to the main bowl, repeat this movement for the middle and right target bowls, and keep repeating this order. They are asked to execute the task as fast as possible.
  Each daily training will consist of three rounds separated by two 5-minute breaks. Each round will consist of four consecutive sessions (for each session: 2-minute training followed by a 30-second break). The training will last for a total of 21 days.
  Arms: the no-RAS group

SUMMARY:
The goal of this clinical trial is to examine effects of training involving rhythmic auditory stimulation (RAS) on upper-limb movements and functions in patients with Parkinson's disease (PD).

This study employed a 21-day randomized controlled trial design to evaluate the efficacy of upper-limb training involving RAS on upper-limb function and neural activity in PD patients. The RAS group showed sustained improvements at one-month follow-up.

DETAILED DESCRIPTION:
This study employed a randomized controlled trial design. We randomly assigned PD patients into either the RAS group (experimental) or the noRAS group (control). Both groups underwent a 21-day training program (40 minutes per session, one session daily), with the only difference being the presence or absence of RAS. Assessments were conducted at five time points: baseline (T1), day 8 (T2), day 15 (T3), post-intervention (T4), and one-month follow-up (T5). Behavioral assessments were performed at all time points, while EEG recordings were only conducted at baseline (T1) and post-intervention (T4). All assessments and training sessions were scheduled during participants' medication 'on' state (1-2 hours after medication intake) to ensure consistency and optimal motor function.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD diagnosed by a neurologist based on the Movement Disorders Society clinical diagnostic criteria;
* the Hoehn and Yahr stage is 2 or 3, meaning that bilateral movement problems or combination with mild postural instability;
* a score of Montreal Cognitive Assessment is equal to or higher than 21 to ensure that they understand experimental instructions;
* a score of Edinburgh Handedness Inventory is above 60 to ensure that they are right-handed;
* types and doses of medications remain unchanged in the past month right before participation.

Exclusion Criteria:

* the presence of medical conditions or diseases that may affect hand movements, vision, or hearing based on self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The box and block test (BBT) | Baseline (T1). Before the training. BBT requires 8-10 minutes to administer.
  BBT is used to measure manual dexterity as well as upper-limb movement speed. It is a 53.7* 25.4 cm box separated into two compartments by a 15.2 cm high erected partition, with 150 blocks in each compartment. Starting from the dominant hand, patients will be asked to move the blocks one by one from the compartment on the hand side to the opposite side (e.g., move the blocks from the right compartment to the left compartment for the right hand test). Patients should move the blocks with their arms raised and crossed over the partition. They have one minute to move the blocks as fast as possible. The score of BBT for each hand is the quantity of blocks transferred between compartments in one minute. A higher score indicates faster upper-limb movements and better dexterity. For the elderly, the BBT has high test-retest reliability (intraclass correlation coefficient of 0.89 to 0.97) and construct validity.
The box and block test (BBT) | Day 8 (T2). During the training. BBT requires 8-10 minutes to administer.
  BBT is used to measure manual dexterity as well as upper-limb movement speed. It is a 53.7* 25.4 cm box separated into two compartments by a 15.2 cm high erected partition, with 150 blocks in each compartment. Starting from the dominant hand, patients will be asked to move the blocks one by one from the compartment on the hand side to the opposite side (e.g., move the blocks from the right compartment to the left compartment for the right hand test). Patients should move the blocks with their arms raised and crossed over the partition. They have one minute to move the blocks as fast as possible. The score of BBT for each hand is the quantity of blocks transferred between compartments in one minute. A higher score indicates faster upper-limb movements and better dexterity. For the elderly, the BBT has high test-retest reliability (intraclass correlation coefficient of 0.89 to 0.97) and construct validity.
The box and block test (BBT) | Day 15 (T3). During the training. BBT requires 8-10 minutes to administer.
  BBT is used to measure manual dexterity as well as upper-limb movement speed. It is a 53.7* 25.4 cm box separated into two compartments by a 15.2 cm high erected partition, with 150 blocks in each compartment. Starting from the dominant hand, patients will be asked to move the blocks one by one from the compartment on the hand side to the opposite side (e.g., move the blocks from the right compartment to the left compartment for the right hand test). Patients should move the blocks with their arms raised and crossed over the partition. They have one minute to move the blocks as fast as possible. The score of BBT for each hand is the quantity of blocks transferred between compartments in one minute. A higher score indicates faster upper-limb movements and better dexterity. For the elderly, the BBT has high test-retest reliability (intraclass correlation coefficient of 0.89 to 0.97) and construct validity.
The box and block test (BBT) | Post-intervention (T4). BBT requires 8-10 minutes to administer.
  BBT is used to measure manual dexterity as well as upper-limb movement speed. It is a 53.7* 25.4 cm box separated into two compartments by a 15.2 cm high erected partition, with 150 blocks in each compartment. Starting from the dominant hand, patients will be asked to move the blocks one by one from the compartment on the hand side to the opposite side (e.g., move the blocks from the right compartment to the left compartment for the right hand test). Patients should move the blocks with their arms raised and crossed over the partition. They have one minute to move the blocks as fast as possible. The score of BBT for each hand is the quantity of blocks transferred between compartments in one minute. A higher score indicates faster upper-limb movements and better dexterity. For the elderly, the BBT has high test-retest reliability (intraclass correlation coefficient of 0.89 to 0.97) and construct validity.
The box and block test (BBT) | One-month follow-up (T5). BBT requires 8-10 minutes to administer.
  BBT is used to measure manual dexterity as well as upper-limb movement speed. It is a 53.7* 25.4 cm box separated into two compartments by a 15.2 cm high erected partition, with 150 blocks in each compartment. Starting from the dominant hand, patients will be asked to move the blocks one by one from the compartment on the hand side to the opposite side (e.g., move the blocks from the right compartment to the left compartment for the right hand test). Patients should move the blocks with their arms raised and crossed over the partition. They have one minute to move the blocks as fast as possible. The score of BBT for each hand is the quantity of blocks transferred between compartments in one minute. A higher score indicates faster upper-limb movements and better dexterity. For the elderly, the BBT has high test-retest reliability (intraclass correlation coefficient of 0.89 to 0.97) and construct validity.
The Jebsen hand function test (JHFT) | Baseline (T1). Before the training. JHFT takes approximately 15 minutes to administer.
  JHFT is used to assess unimanual hand function when examinees perform daily activities. Seven items are included in JHFT: writing, turning cards, picking up small objects, simulated feeding, stacking checkers, moving large light objects, and moving large heavy objects. Considering that the patients are Chinese speakers, it is not appropriate to do English writing. According to a previous study conducted in Chinese cultures, the JHFT could be modified through excluding the writing item to avoid cultural influences on scores. The score for each item is the completion time. The less time a patient takes, the better hand function s/he has. The JHFT has excellent test-retest reliability (intraclass correlation coefficients of 0.89 to 0.97) for PD patients.
The Jebsen hand function test (JHFT) | Day 8 (T2). During the training. JHFT takes approximately 15 minutes to administer.
  JHFT is used to assess unimanual hand function when examinees perform daily activities. Seven items are included in JHFT: writing, turning cards, picking up small objects, simulated feeding, stacking checkers, moving large light objects, and moving large heavy objects. Considering that the patients are Chinese speakers, it is not appropriate to do English writing. According to a previous study conducted in Chinese cultures, the JHFT could be modified through excluding the writing item to avoid cultural influences on scores. The score for each item is the completion time. The less time a patient takes, the better hand function s/he has. The JHFT has excellent test-retest reliability (intraclass correlation coefficients of 0.89 to 0.97) for PD patients.
The Jebsen hand function test (JHFT) | Day 15 (T3). During the training. JHFT takes approximately 15 minutes to administer.
  JHFT is used to assess unimanual hand function when examinees perform daily activities. Seven items are included in JHFT: writing, turning cards, picking up small objects, simulated feeding, stacking checkers, moving large light objects, and moving large heavy objects. Considering that the patients are Chinese speakers, it is not appropriate to do English writing. According to a previous study conducted in Chinese cultures, the JHFT could be modified through excluding the writing item to avoid cultural influences on scores. The score for each item is the completion time. The less time a patient takes, the better hand function s/he has. The JHFT has excellent test-retest reliability (intraclass correlation coefficients of 0.89 to 0.97) for PD patients.
The Jebsen hand function test (JHFT) | Post-intervention (T4). JHFT takes approximately 15 minutes to administer.
  JHFT is used to assess unimanual hand function when examinees perform daily activities. Seven items are included in JHFT: writing, turning cards, picking up small objects, simulated feeding, stacking checkers, moving large light objects, and moving large heavy objects. Considering that the patients are Chinese speakers, it is not appropriate to do English writing. According to a previous study conducted in Chinese cultures, the JHFT could be modified through excluding the writing item to avoid cultural influences on scores. The score for each item is the completion time. The less time a patient takes, the better hand function s/he has. The JHFT has excellent test-retest reliability (intraclass correlation coefficients of 0.89 to 0.97) for PD patients.
The Jebsen hand function test (JHFT) | One-month follow-up (T5). JHFT takes approximately 15 minutes to administer.
  JHFT is used to assess unimanual hand function when examinees perform daily activities. Seven items are included in JHFT: writing, turning cards, picking up small objects, simulated feeding, stacking checkers, moving large light objects, and moving large heavy objects. Considering that the patients are Chinese speakers, it is not appropriate to do English writing. According to a previous study conducted in Chinese cultures, the JHFT could be modified through excluding the writing item to avoid cultural influences on scores. The score for each item is the completion time. The less time a patient takes, the better hand function s/he has. The JHFT has excellent test-retest reliability (intraclass correlation coefficients of 0.89 to 0.97) for PD patients.
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale motor section (MDS-UPDRS III) | Baseline (T1). Before the training. MDS-UPDRS III takes approximately 15 minutes to administer.
  The MDS-UPDRS evaluates various aspects of PD, including four parts: subjective non-motor experiences of daily living, subjective motor experiences of daily living, motor examination of the motor signs of PD, and motor complications based on historical and objective information. The scale is widely used in clinical settings as well as in research. We calculated the score of MDS-UPDRS Ⅲ, which is the motor examination of the motor signs, to assess the severity of bradykinesia.
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale motor section (MDS-UPDRS III) | Post-intervention (T4). MDS-UPDRS III takes approximately 15 minutes to administer.
  The MDS-UPDRS evaluates various aspects of PD, including four parts: subjective non-motor experiences of daily living, subjective motor experiences of daily living, motor examination of the motor signs of PD, and motor complications based on historical and objective information. The scale is widely used in clinical settings as well as in research. We calculated the score of MDS-UPDRS Ⅲ, which is the motor examination of the motor signs, to assess the severity of bradykinesia.
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale motor section (MDS-UPDRS III) | One-month follow-up (T5). MDS-UPDRS III takes approximately 15 minutes to administer.
  The MDS-UPDRS evaluates various aspects of PD, including four parts: subjective non-motor experiences of daily living, subjective motor experiences of daily living, motor examination of the motor signs of PD, and motor complications based on historical and objective information. The scale is widely used in clinical settings as well as in research. We calculated the score of MDS-UPDRS Ⅲ, which is the motor examination of the motor signs, to assess the severity of bradykinesia.
The Nine-Hole Peg Test (NHPT) | Baseline (T1). Before the training. Before the training. NHPT takes approximately 5 minutes to administer.
  The NHPT is widely used measure of hand dexterity in a broad range of ages and population. The NHPT requires participants to quickly pick up nine small pegs from a concave receptacle, place them into holes on a board as fast as possible, and then move them back to the receptacle. The total time has been recorded as the result of NHPT, the less time taken indicate better hand dexterity. It has a high test-retest reliability for both hand (intraclass correlation coefficients of 0.88 to 0.91) and construct validity in PD population.
The Nine-Hole Peg Test (NHPT) | Day 8 (T2). During the training. NHPT takes approximately 5 minutes to administer.
  The NHPT is widely used measure of hand dexterity in a broad range of ages and population. The NHPT requires participants to quickly pick up nine small pegs from a concave receptacle, place them into holes on a board as fast as possible, and then move them back to the receptacle. The total time has been recorded as the result of NHPT, the less time taken indicate better hand dexterity. It has a high test-retest reliability for both hand (intraclass correlation coefficients of 0.88 to 0.91) and construct validity in PD population.
The Nine-Hole Peg Test (NHPT) | Day 15 (T3). During the training. NHPT takes approximately 5 minutes to administer.
  The NHPT is widely used measure of hand dexterity in a broad range of ages and population. The NHPT requires participants to quickly pick up nine small pegs from a concave receptacle, place them into holes on a board as fast as possible, and then move them back to the receptacle. The total time has been recorded as the result of NHPT, the less time taken indicate better hand dexterity. It has a high test-retest reliability for both hand (intraclass correlation coefficients of 0.88 to 0.91) and construct validity in PD population.
The Nine-Hole Peg Test (NHPT) | Post-intervention (T4). NHPT takes approximately 5 minutes to administer.
  The NHPT is widely used measure of hand dexterity in a broad range of ages and population. The NHPT requires participants to quickly pick up nine small pegs from a concave receptacle, place them into holes on a board as fast as possible, and then move them back to the receptacle. The total time has been recorded as the result of NHPT, the less time taken indicate better hand dexterity. It has a high test-retest reliability for both hand (intraclass correlation coefficients of 0.88 to 0.91) and construct validity in PD population.
The Nine-Hole Peg Test (NHPT) | One-month follow-up (T5). NHPT takes approximately 5 minutes to administer.
  The NHPT is widely used measure of hand dexterity in a broad range of ages and population. The NHPT requires participants to quickly pick up nine small pegs from a concave receptacle, place them into holes on a board as fast as possible, and then move them back to the receptacle. The total time has been recorded as the result of NHPT, the less time taken indicate better hand dexterity. It has a high test-retest reliability for both hand (intraclass correlation coefficients of 0.88 to 0.91) and construct validity in PD population.

SECONDARY OUTCOMES:
Electroencephalography (EEG) | Baseline (T1). Before the training. It takes about 20 minutes to complete all the EEG recording procedures, including setup and removal.
  EEG recordings were conducted using a clinical-grade Nicolet Monitor system (Natus Medical Incorporated, USA). The system features comprehensive neurophysiological monitoring capabilities with high signal-to-noise ratio and stable recording characteristics. We employed a standard 19-electrode montage following the international 10-20 system, ensuring precise and reproducible electrode positioning based on anatomical landmarks.
Electroencephalography (EEG) | Post-intervention (T4). It takes about 20 minutes to complete all the EEG recording procedures, including setup and removal.
  EEG recordings were conducted using a clinical-grade Nicolet Monitor system (Natus Medical Incorporated, USA). The system features comprehensive neurophysiological monitoring capabilities with high signal-to-noise ratio and stable recording characteristics. We employed a standard 19-electrode montage following the international 10-20 system, ensuring precise and reproducible electrode positioning based on anatomical landmarks.

CONTACTS AND LOCATIONS:
Overall Officials: Wei FAN (PhD student), MSc, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bengtsson SL, Ullen F, Ehrsson HH, Hashimoto T, Kito T, Naito E, Forssberg H, Sadato N. Listening to rhythms activates motor and premotor cortices. Cortex. 2009 Jan;45(1):62-71. doi: 10.1016/j.cortex.2008.07.002. Epub 2008 Oct 30. PMID 19041965
- [Background] Braunlich K, Seger CA, Jentink KG, Buard I, Kluger BM, Thaut MH. Rhythmic auditory cues shape neural network recruitment in Parkinson's disease during repetitive motor behavior. Eur J Neurosci. 2019 Mar;49(6):849-858. doi: 10.1111/ejn.14227. Epub 2018 Dec 3. PMID 30375083
- [Background] Buard I, Dewispelaere WB, Thaut M, Kluger BM. Preliminary Neurophysiological Evidence of Altered Cortical Activity and Connectivity With Neurologic Music Therapy in Parkinson's Disease. Front Neurosci. 2019 Feb 19;13:105. doi: 10.3389/fnins.2019.00105. eCollection 2019. PMID 30837830
- [Background] Cahn DA, Sullivan EV, Shear PK, Pfefferbaum A, Heit G, Silverberg G. Differential contributions of cognitive and motor component processes to physical and instrumental activities of daily living in Parkinson's disease. Arch Clin Neuropsychol. 1998 Oct;13(7):575-83. PMID 14590618
- [Background] Chen JL, Penhune VB, Zatorre RJ. Listening to musical rhythms recruits motor regions of the brain. Cereb Cortex. 2008 Dec;18(12):2844-54. doi: 10.1093/cercor/bhn042. Epub 2008 Apr 3. PMID 18388350
- [Background] Dalrymple-Alford JC, MacAskill MR, Nakas CT, Livingston L, Graham C, Crucian GP, Melzer TR, Kirwan J, Keenan R, Wells S, Porter RJ, Watts R, Anderson TJ. The MoCA: well-suited screen for cognitive impairment in Parkinson disease. Neurology. 2010 Nov 9;75(19):1717-25. doi: 10.1212/WNL.0b013e3181fc29c9. PMID 21060094
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Dong VA, Fong KN, Chen YF, Tseng SS, Wong LM. 'Remind-to-move' treatment versus constraint-induced movement therapy for children with hemiplegic cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2017 Feb;59(2):160-167. doi: 10.1111/dmcn.13216. Epub 2016 Aug 9. PMID 27503605
- [Background] Fan W, Li J, Wei W, Xiao SH, Liao ZJ, Wang SM, Fong KNK. Effects of rhythmic auditory stimulation on upper-limb movements in patients with Parkinson's disease. Parkinsonism Relat Disord. 2022 Aug;101:27-30. doi: 10.1016/j.parkreldis.2022.06.020. Epub 2022 Jun 23. PMID 35763906
- [Background] Gale JT, Amirnovin R, Williams ZM, Flaherty AW, Eskandar EN. From symphony to cacophony: pathophysiology of the human basal ganglia in Parkinson disease. Neurosci Biobehav Rev. 2008;32(3):378-87. doi: 10.1016/j.neubiorev.2006.11.005. Epub 2007 Apr 26. PMID 17466375
- [Background] Ghai S, Ghai I, Schmitz G, Effenberg AO. Effect of rhythmic auditory cueing on parkinsonian gait: A systematic review and meta-analysis. Sci Rep. 2018 Jan 11;8(1):506. doi: 10.1038/s41598-017-16232-5. PMID 29323122
- [Background] Grahn JA, Rowe JB. Feeling the beat: premotor and striatal interactions in musicians and nonmusicians during beat perception. J Neurosci. 2009 Jun 10;29(23):7540-8. doi: 10.1523/JNEUROSCI.2018-08.2009. PMID 19515922
- [Background] Jastrzebowska MA, Marquis R, Melie-Garcia L, Lutti A, Kherif F, Herzog MH, Draganski B. Dopaminergic modulation of motor network compensatory mechanisms in Parkinson's disease. Hum Brain Mapp. 2019 Oct 15;40(15):4397-4416. doi: 10.1002/hbm.24710. Epub 2019 Jul 10. PMID 31291039
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Background] Koshimori Y, Thaut MH. Future perspectives on neural mechanisms underlying rhythm and music based neurorehabilitation in Parkinson's disease. Ageing Res Rev. 2018 Nov;47:133-139. doi: 10.1016/j.arr.2018.07.001. Epub 2018 Jul 10. PMID 30005957
- [Background] Kraft E, Loichinger W, Diepers M, Lule D, Schwarz J, Ludolph AC, Storch A. Levodopa-induced striatal activation in Parkinson's disease: a functional MRI study. Parkinsonism Relat Disord. 2009 Sep;15(8):558-63. doi: 10.1016/j.parkreldis.2009.02.005. Epub 2009 May 20. PMID 19467909
- [Background] Leuk JSP, Low LLN, Teo WP. An Overview of Acoustic-Based Interventions to Improve Motor Symptoms in Parkinson's Disease. Front Aging Neurosci. 2020 Aug 14;12:243. doi: 10.3389/fnagi.2020.00243. eCollection 2020. PMID 32922283
- [Background] Mak MK, Lau ET, Tam VW, Woo CW, Yuen SK. Use of Jebsen Taylor Hand Function Test in evaluating the hand dexterity in people with Parkinson's disease. J Hand Ther. 2015 Oct-Dec;28(4):389-94; quiz 395. doi: 10.1016/j.jht.2015.05.002. Epub 2015 May 18. PMID 26227308
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Muslimovic D, Post B, Speelman JD, Schmand B, de Haan RJ; CARPA Study Group. Determinants of disability and quality of life in mild to moderate Parkinson disease. Neurology. 2008 Jun 3;70(23):2241-7. doi: 10.1212/01.wnl.0000313835.33830.80. PMID 18519873
- [Background] Ni M, Hazzard JB, Signorile JF, Luca C. Exercise Guidelines for Gait Function in Parkinson's Disease: A Systematic Review and Meta-analysis. Neurorehabil Neural Repair. 2018 Oct;32(10):872-886. doi: 10.1177/1545968318801558. Epub 2018 Sep 28. PMID 30265211
- [Background] Nombela C, Hughes LE, Owen AM, Grahn JA. Into the groove: can rhythm influence Parkinson's disease? Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2564-70. doi: 10.1016/j.neubiorev.2013.08.003. Epub 2013 Sep 3. PMID 24012774
- [Background] Nonnekes J, Timmer MH, de Vries NM, Rascol O, Helmich RC, Bloem BR. Unmasking levodopa resistance in Parkinson's disease. Mov Disord. 2016 Nov;31(11):1602-1609. doi: 10.1002/mds.26712. Epub 2016 Jul 19. PMID 27430479
- [Background] Radhakrishnan DM, Goyal V. Parkinson's disease: A review. Neurol India. 2018 Mar-Apr;66(Supplement):S26-S35. doi: 10.4103/0028-3886.226451. PMID 29503325
- [Background] Rajiah K, Maharajan MK, Yeen SJ, Lew S. Quality of Life and Caregivers' Burden of Parkinson's Disease. Neuroepidemiology. 2017;48(3-4):131-137. doi: 10.1159/000479031. Epub 2017 Jul 21. PMID 28728161
- [Background] Redgrave P, Rodriguez M, Smith Y, Rodriguez-Oroz MC, Lehericy S, Bergman H, Agid Y, DeLong MR, Obeso JA. Goal-directed and habitual control in the basal ganglia: implications for Parkinson's disease. Nat Rev Neurosci. 2010 Nov;11(11):760-72. doi: 10.1038/nrn2915. Epub 2010 Oct 14. PMID 20944662
- [Background] Schaffert N, Janzen TB, Mattes K, Thaut MH. A Review on the Relationship Between Sound and Movement in Sports and Rehabilitation. Front Psychol. 2019 Feb 12;10:244. doi: 10.3389/fpsyg.2019.00244. eCollection 2019. PMID 30809175
- [Background] Sian J, Gerlach M, Youdim MB, Riederer P. Parkinson's disease: a major hypokinetic basal ganglia disorder. J Neural Transm (Vienna). 1999;106(5-6):443-76. doi: 10.1007/s007020050171. PMID 10443550
- [Background] Thaut MH, McIntosh GC, Rice RR, Miller RA, Rathbun J, Brault JM. Rhythmic auditory stimulation in gait training for Parkinson's disease patients. Mov Disord. 1996 Mar;11(2):193-200. doi: 10.1002/mds.870110213. PMID 8684391
- [Background] Thaut MH, McIntosh GC, Hoemberg V. Neurobiological foundations of neurologic music therapy: rhythmic entrainment and the motor system. Front Psychol. 2015 Feb 18;5:1185. doi: 10.3389/fpsyg.2014.01185. eCollection 2014. PMID 25774137
- [Background] Vitorio R, Stuart S, Gobbi LTB, Rochester L, Alcock L, Pantall A. Reduced Gait Variability and Enhanced Brain Activity in Older Adults With Auditory Cues: A Functional Near-Infrared Spectroscopy Study. Neurorehabil Neural Repair. 2018 Nov;32(11):976-987. doi: 10.1177/1545968318805159. PMID 30411674
- [Background] Vorovenci RJ, Biundo R, Antonini A. Therapy-resistant symptoms in Parkinson's disease. J Neural Transm (Vienna). 2016 Jan;123(1):19-30. doi: 10.1007/s00702-015-1463-8. Epub 2015 Sep 26. PMID 26410626
- [Background] Yang N, Waddington G, Adams R, Han J. Translation, cultural adaption, and test-retest reliability of Chinese versions of the Edinburgh Handedness Inventory and Waterloo Footedness Questionnaire. Laterality. 2018 May;23(3):255-273. doi: 10.1080/1357650X.2017.1357728. Epub 2017 Jul 31. PMID 28756732
- [Derived] Fan W, Fong KNK, Wang SM. Effects of training involving patterned sensory enhancement on improving upper-limb movements in patients with Parkinson's disease: protocol of a randomised controlled trial. BMJ Open. 2023 Jul 12;13(7):e072416. doi: 10.1136/bmjopen-2023-072416. PMID 37438071